CLINICAL TRIAL: NCT00782665
Title: Myometrial Biopsy for the Detection of Infection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Woman's Hospital of Texas (Other)
Responsible Party: Sebastian Faro, MD, PhD, The Woman's Hospital of Texas
Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10012008Faro
Record Dates: First submitted 2008-10-28; First posted 2008-10-31 (Estimated); Last update posted 2008-10-31 (Estimated); Status verified 2008-10

CONDITIONS: Infection
Keywords: postoperative; infection; c-section
MeSH Terms: conditions — Infections | interventions — Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Active Comparator): Patients who have labored and subsequently delivered by cesarean section
  Interventions: Procedure: Biopsy
- 2 (Placebo Comparator): Patients who electively select cesarean section
  Interventions: Procedure: Biopsy

INTERVENTIONS:
Procedure: Biopsy — 1 centimeter x 1/2 centimeter piece cut from uterus

SUMMARY:
This study is designed to demonstrate that women in labor become infected without exhibiting any clinical signs or symptoms of infection.

DETAILED DESCRIPTION:
The infection is a dynamic process probably beginning shortly after the onset of labor. This process continues and is enhanced during active uterine contractions, which result in bacteria from the vagina being drawn up into the uterine cavity. During labor, bacterial colonization of the amniotic fluid, the decidua, and even the fetus can occur, resulting in infection of the mother and the fetus.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be afebrile throughout labor.
2. Amniotic fluid must be not purulent; presence of meconium is not an exclusion.
3. Patients undergoing an elective cesarean section.
4. Patients who have labored with intact or ruptured amniotic membranes.

Exclusion Criteria:

1. Patient with a temperature of ≥ 100.4o F.
2. White blood cell count ≥ 24,000.
3. Suspicion of chorioamnionitis.
4. Suspicion of a urinary tract infection.
5. Presence of diarrhea (defined > 4 liquid stools in a 24 hour period).
6. Patient currently taking therapeutic antibiotics.

Ages: 18 Years to 48 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1000 (Estimated)
Dates: Start 2008-07; Primary Completion 2010-06 (Estimated); Study Completion 2010-07 (Estimated)

PRIMARY OUTCOMES:
Postoperative infection following rupture of amniotic membranes | Amount of time it takes to obtain culture result

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian Faro, MD, PhD, Principal Investigator — The Woman's Hospital of Texas
Locations (1):
- The Woman's Hospital of Texas, Houston, Texas, United States